CLINICAL TRIAL: NCT02622633
Title: Epidural Stimulation for Resistant Depression Treatment: A Randomized Double Blind Clinical Trial
Brief Title: Epidural Stimulation for Resistant Depression Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Monique Gomes da Silva Scalco, Principal Investigator, University of Brasilia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 40803214.2.0000.0033
Record Dates: First submitted 2015-11-30; First posted 2015-12-04 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation (Experimental): One week after implantation of the device, participants randomized in this arm will receive continuous magnetic stimulation of high frequency (50Hz) with epidural electrode for 12 weeks. And then, the epidural electrode will be turned off for more 12 weeks in a crossover fashion.
  Interventions: Device: Epidural Electrode
- Sham Stimulation (Sham Comparator): One week after implantation of the device, participants randomized in this arm will receive sham stimulation for 12 weeks and then continuous magnetic stimulation with epidural electrode of high frequency (50Hz) stimulation for more 12 weeks.
  Interventions: Device: Epidural Electrode

INTERVENTIONS:
Device: Epidural Electrode — Epidural electrode of high frequency (50Hz) stimulation in the dorsolateral prefrontal cortex.

SUMMARY:
This study aims to analyze the effectiveness and feasibility of using an implantable system that provides epidural electrical stimulation directly to the left prefrontal dorsolateral cortex (Brodmann area 9/46) in patients with chronic and refractory Depressive Disorder Major.

DETAILED DESCRIPTION:
Exploratory Objectives

To analyze the hypothetical advantages of epidural cortical stimulation compare to less invasive method of transcranial magnetic stimulation:

* Surgical implantation of stimulating electrodes can lead to a more powerful, consistent and accurate form of stimulation to the cortex, one of the main concerns associated with the variability observed in studies of transcranial magnetic stimulation.
* A definitive system for the implantation could also overcome another disadvantage of transcranial magnetic stimulation therapy, the need of repetitive treatment period of several weeks, and the need for maintenance sessions.
* To achieve remission of depressive symptoms by promoting improved quality of life and reducing the risk of suicide.
* To improve patient adherence to the treatment by the establishment of a permanent system.

Sample:

Patients will be selected from outpatient clinics and psychiatric wards of specialized services in Distrito Federal, Brasília, Brazil. These patients will be included in a specific outpatient affective disorders at the University Hospital of Brasília. Those patients with major depressive disorder considered untreatable by conventional methods:

1. The inclusion in this study requires that patients meet the criteria for recurrent Major Depressive Disorder according to the Diagnostic and Statistical Manual - V (recurrent Major Depressive Disorder without psychotic features), being in a current depressive episode lasting at least two years or have produced at least four episodes of major depression, along with the current episode lasting at least one year. All individuals must be adults, women can not be pregnant and must be submitted to contraceptive therapy.
2. Subjects must have failed to respond to at least four different trials with antidepressant at therapeutic doses for a period of at least six weeks, associated with specific psychotherapy during this period and/or use of electrochemotherapy or vagal nerve stimulation . The medication treatment for depression used at the moment of selection should remain unchanged for at least eight weeks after implantation and will not change during the study period. Possible needs therapeutic adjustments during the study will be managed with changes in parameter magnetic stimulation.
3. Patients should score at least 20 points on the Hamilton Rating Scale (Hamilton Depression Rating Scale-28 (HDRS)
4. Exclusion criteria:

   1. Pregnancy;
   2. Preexisting neurological disease including epilepsy;
   3. Other psychiatric disorders except for anxiety disorders
   4. Less than 24 Mini-Mental or any other cognitive disorder;
   5. Being with serious suicidal ideation.
   6. Medical conditions that preclude surgery as judgment of the research team.

Rating Scales:

1. Rating Scale Hamilton Depression (HAM-D), the 28 items: assessment of severity of symptoms in depressed patients with primary depressive illness and monitoring changes due to treatment.
2. Depression Scale Montgomery-Asberg Depression Rating Scale (MADRS), specific evaluation of clinical changes in depressed patients during treatment.
3. Scale of the SF-36, evaluates subjectively the individual's perception regarding their own health.
4. Side Effects Scale (UKU- Ugvalg is Kliniske Undersgelser): detailed scale for assessment of drug side effects comprising the following four groups of side effects: psychic, neurological, autonomic and others.

Procedures:

Selected patients will undergo surgical implant procedure performed at the Surgical Center of the University Hospital of Brasília (HUB). The implant will be done by a specialist neurosurgeon in the treatment of functional disorders and in implantation of epidural electrodes for other pathologies. The procedure will be done using neuronavigation and the implant material is already acquired by the neurosurgery unit of HUB by direct import.

Risks associated with surgery:

* Risk of system infection: 3%
* Risk of surgical hematoma: 0.2%
* Risk of death: 0.1%
* Risk of neurological sequelae: 0.1%

Timeline:

* Patients will be selected in outpatient Psychiatry, University Hospital of Brasilia. This clinic will be conducted by psychiatrists and psychiatry residents and it will be specific to patients with major depression and clinical management difficult.
* After obtaining informed consent and informed consent and resolved all questions from participants about the research, patients who agree to participate in the study will undergo a general physical examination, neurological evaluation, EEG assessment and neuropsychological assessment. Depression severity will be assessed by the Hamilton scale (HAM-17). Secondary measures of depression severity will be assessed with the Depression Scale Montgomery-Asberg Depression Rating Scale (MADRS) and the Scale of the SF-36.
* Imaging exam (Positrons Emission Tomography - PET) pre-procedure will be performed.
* Psychiatric diagnoses are excluded by structured interview, including history of previous treatment with the respective drugs used, length of treatment and therapeutic response.
* To the patients who meet inclusion criteria of this research will be offered the possibility of the definitive implant with epidural electrode.
* Realization of imaging examination for surgical planning and anatomical and functional brain assessment.
* In case of agreement, participants who meet inclusion criteria will be forwarded to the implantation of an epidural electrode at the HUB by a trained neurosurgeon in psychosurgery.
* One week after implantation of the device, participants will be randomized in order to receive continuous magnetic stimulation of high frequency (50Hz) stimulation or sham stimulation (placebo) in the first eight weeks of the study. After eight weeks, patients randomized to receive sham stimulation will receive stimulation 50Hz also for eight weeks. At no time participants will be informed of which are part of the research group.
* Completed eight weeks of continuous stimulation at 50 Hz (in the eighth week of the subjects with stimulation at 50Hz and sixteenth week for those who made the first eight weeks of sham stimulation), patients enter into adaptive protocol based on individual response.
* New imaging test (PET) will be held at or after 28 weeks of treatment response criteria achieved, whichever comes first.
* Patients will be reassessed every two weeks for a period of 16 weeks with reapplication of HAM-17 and MADRS. During these reassessments will also be investigated possible adverse effects and patients will have their devices checked stimulation.
* The results will then be subjected to statistical analysis in order to verify the effectiveness of the method.

ELIGIBILITY:
Inclusion Criteria:

1. The inclusion in this study requires that patients meet the criteria for recurrent Major Depressive Disorder according to the DSM V (recurrent Major Depressive Disorder without psychotic features), being in a current depressive episode lasting at least two years or have produced at least four episodes of major depression, along with the current episode lasting at least one year. All individuals must be adults, women can not be pregnant and must be submitted to contraceptive therapy
2. Subjects must have failed to respond to at least four different trials with antidepressant at therapeutic doses for a period of at least six weeks, associated with specific psychotherapy during this period and/or use of ECT or VNS. The medication treatment for depression used at the moment of selection should remain unchanged for at least eight weeks after implantation and will not change during the study period. Possible needs therapeutic adjustments during the study will be managed with changes in parameter magnetic stimulation
3. Patients should score at least 20 points on the Hamilton Rating Scale (Hamilton Depression Rating Scale-28 (HDRS))

Exclusion Criteria:

1. Pregnancy
2. Preexisting neurological disease including epilepsy
3. Other psychiatric disorders except for anxiety disorders
4. Less than 24 Mini-Mental or any other cognitive disorder
5. Being with serious suicidal ideation
6. Medical conditions that preclude surgery as judgment of the research team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Rating Scale Hamilton Depression | baseline - 12 weeks - 26 weeks
  assessment of severity of symptoms in depressed patients with primary depressive illness and monitoring changes due to treatment

SECONDARY OUTCOMES:
Change in Depression Scale Montgomery-Asberg Depression Rating Scale | Baseline - 12 weeks -26 weeks
Change in Scale of the SF-36 | Baseline - 12 weeks -26 weeks
  evaluates subjectively the individual's perception regarding their own health
Frequency of Side Effects Scale - (UKU- Ugvalg is Kliniske Undersgelser) | Baseline - 12 weeks - 26 weeks
  detailed scale for assessment of drug side effects comprising the following four groups of side effects: psychic, neurological, autonomic and others

CONTACTS AND LOCATIONS:
Locations (1):
- Rivadavio Amorim, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The data will be available in the institution - Brasilia University.